CLINICAL TRIAL: NCT03298542
Title: A Phase 1b Study to Evaluate SIMPONI (Golimumab) Therapy in Children, Adolescents and Young Adults With Pre-Symptomatic Type 1 Diabetes
Brief Title: A Study to Evaluate SIMPONI (Golimumab) Therapy in Children, Adolescents and Young Adults With Pre-Symptomatic Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108354; 2017-000225-12 (EudraCT Number); CNTO148DML1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-09-15; First posted 2017-10-02 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pre-Symptomatic Type 1 Diabetes
MeSH Terms: interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Golimumab (Experimental): Participants will receive subcutaneous (SC) golimumab for 26 weeks, where doses will be based on weight and/or body surface area.
  Interventions: Drug: Golimumab
- Group 2: Placebo (Placebo Comparator): Participants will receive a SC matching placebo to golimumab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Golimumab — Participants will receive subcutaneous golimumab for 26 weeks, where doses will be based on weight and/or body surface area.
  Other Names: SIMPONI
  Arms: Group 1: Golimumab
Drug: Placebo — Matching placebo to golimumab.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of golimumab in children, adolescents, and young adults with pre-symptomatic stage 2 type 1 diabetes mellitus (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Is positive for at least 2 of the following diabetes-related autoantibodies obtained at study screening: Glutamic acid decarboxylase-65 (GAD-65) Autoantibodies, Insulinoma-associated 2 Autoantibodies (IA-2A), Zinc Transporter-8 (ZnT8), Islet Cell Cytoplasmic Autoantibodies (ICA), or Insulin Autoantibodies (IAA). Participants with a confirmed documented history of at least 2 positive diabetes-related autoantibodies but who screen positive on only 1 autoantibody are considered to have met this criteria
* Has a plasma glucose of 7.8 to 11.0 millimoles per liter (mmol/L) (140 to 199 milligrams per deciliter (mg/dL)) at the 120-minute timepoint of a 2-hour(h)-oral glucose tolerance test (OGTT), OR have a plasma glucose of greater than (>) 200 mg/dL (> 11.1 mmol/L) at the 30, 60, or 90 minute timepoint of a 2h-OGTT OR have a hemoglobin A1c (HbA1c) greater than or equal to (>=) 5.7 percent (%) but less than (<) 6.5% ([>=] 39 to <48 millimoles per moles [mmol/mol]) evaluated at screening
* Is medically stable on the basis of physical examination, medical history, laboratory results, and vital signs performed at screening
* If a woman of childbearing potential must have a negative highly sensitive serum test (beta-human chorionic gonadotropin) at screening and a negative urine pregnancy test at the Week 0 visit
* Must be up-to-date or have initiated catch up vaccines with routine age-appropriate immunizations and have received vaccines, or at least initiated vaccine series and have a completion plan, that are recommended for immune suppressed individuals according to current local recommendations before the first dose of study treatment

Exclusion Criteria:

* Has a current or prior diagnosis of diabetes mellitus (Type 1, Type 2, or gestational) or meet the metabolic criteria diagnostic of diabetes mellitus obtained at screening including: hemoglobin A1c (HbA1c) greater than or equal to 6.5 (%) (48 mmol/mol), or fasting plasma glucose (>=) 7.0 mmol/L (126 mg/dL) (fasting: no intake >= 8 hours), or plasma glucose >= 11.1 mmol/L (200 mg/dL) 2 hours post OGTT, or random plasma glucose >= 11.1 mmol/L (200 mg/dL) in those with symptoms consistent with hyperglycemia crisis
* Has a presence or history of malignancy
* Has an immune deficiency syndrome (for example, severe combined immunodeficiency syndrome, T-cell deficiency syndromes, B-cell deficiency syndromes, or chronic granulomatous disease), or bone marrow or organ transplantation, or a disease associated with lymphopenia
* Has other autoimmune diseases (for example, rheumatoid arthritis (RA), polyarticular juvenile idiopathic arthritis (pJIA), psoriatic arthritis (PsA), ankylosing spondylitis (AS), multiple sclerosis, celiac disease, systemic lupus erythematosus) excluding clinically stable autoimmune thyroiditis whether treated or untreated
* Has active infections, is prone to infections or has chronic, recurrent or opportunistic infectious disease, including but not limited to, chronic renal infection, chronic chest infection, sinusitis, recurrent urinary tract infection, Pneumocystis carinii, aspergillosis, latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis or an open, draining, or infected non healing skin wound or ulcer
* Has a clinically active infection with Epstein-Barr virus (EBV) or an EBV polymerase chain reaction (PCR) viral load serology of >= 10,000 copies per milliliter (mL) at study screening
* Has a clinically active infection with cytomegalovirus (CMV) or a CMV PCR viral load serology of >= 10,000 copies per mL at study screening
* Is infected with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) or at screening tests positive for HIV, HBV, or HCV
* Has any of the following tuberculosis (TB) screening criteria: a history of latent or active TB prior to screening; signs or symptoms suggestive of active TB upon medical history and/or physical examination; recent close contact (within 3 months) with a person with known or suspected active TB; a positive QuantiFERON-TB test result at screening, the participant should be excluded from the study; a chest radiograph taken within 3 months prior to the first administration of study treatment read by a qualified radiologist consistent with current, active TB or old, inactive TB
* Has a current or prior use of any type and form of exogenous insulin or oral/intravenous (IV) antihyperglycemic treatment
* Has known or suspected intolerance or hypersensitivity to human proteins, antibody fragments, or monoclonal antibodies, including golimumab or its excipients

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 26
Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 52
Percentage of Participants With Treatment-Emergent Infections | Up to Week 26
Percentage of Participants With Treatment-Emergent Infections | Up to Week 52
Percentage of Participants With Study Treatment Injection Site Reactions | Up to Week 26
Number of Participants With Treatment Related AEs and SAEs Reported From Week 52 to Week 78 | Week 52 to Week 78

SECONDARY OUTCOMES:
Serum Concentration of Golimumab | Through Week 52
Incidence of Antibodies to Golimumab | Through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (3):
  - UC Denver-Colorado Barbara Davis Center, University of Colorado SOM Pediatric Endocrinology, Aurora, Colorado
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Finland (3):
  - Oulu University Hosp. Oulu, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Sweden (2):
  - Linkoping University Hospital, Linköping
  - Lund University Hospital/Skåne, Lund/Malmo

REFERENCES:
- See also: Link to results on EudraCT registry. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2017-000225-12/results